CLINICAL TRIAL: NCT00303433
Title: Namenda as Prevention for Post-Operative Delirium
Brief Title: Namenda to Prevent Post-Operative Delirium
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Forest Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RSRB-00012460; NAM-MD-35; NCT00303095 (obsolete NCT alias)
Record Dates: First submitted 2006-03-14; First posted 2006-03-16 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2009-12

CONDITIONS: Delirium; Post-Operative States
Keywords: Prevention; Post-Operative tates; Delirium; Namenda
MeSH Terms: conditions — Delirium | interventions — Memantine

INTERVENTIONS:
Drug: Namenda

SUMMARY:
Post Operative Delirium is a common and serious risk of surgery. Delirium, when it occurs is associated with an increased risk of mortality, increase length of stay, and more adverse outcomes in general, including increased risk of higher level of care required at discharge.

Namenda, which is currently approved for moderate or severe Alzheimer's disease has a unique mechanism of action than other drugs for this condition. It may have the ability to protect the brain from more severe consequences of hypoxia, or hypoglycemia. Hence it is being looked at in this study to see if it can reduce the incidence and/or severity of delirium post-operatively.

DETAILED DESCRIPTION:
Objectives of this double blind placebo-controlled study are to determine the efficacy, safety and tolerability of Namenda in the prevention of post-operative delirium as defined by DSM-IV-TR categories 293.0 Delirium due to medical condition or medications, and 780.09 Delirium NOS. The incidence of post-operative delirium is 10-50% of general surgical cases, depending on the population studied. Delirium is known to affect mortality and morbidity, and increase the length of stay of patients. Hospital mortality estimates in patients with delirium range from 10-65%, estimated to be 2-20 times that of control patients without delirium. Delirium is an independent prognostic determinant of hospital outcomes, including death, new nursing home placements and functional decline. Delirium is an independent marker for increased mortality among older medical inpatients in the 12 months post hospitalization, particularly in those patients without dementia.

Delirium may be better understood by a Multifactorial Model of Delirium, which involves a complex inter-relationship between predisposing Factors/Vulnerability and Precipitating Factors/Insults.

If higher risk factors can be identified, then preventive interventions targeted to these groups may be able to significantly reduce morbitity, possibly mortality, but at minimum improve the quality of life of those patients who otherwise would have gone through such an enormously traumatic and disturbing experience as the psychosis and disorientation of a delirium.

The Academy of Psyhosomatic Medicine Task Force on Mental Disorders in General Medical Practice, found that co-morbid delirium increased hospital length of stay: 100% in general medical inpatients, 114% in elderly patients, 67% in stroke patients, 300% in critical care patients, 27% in cardiac surgery patients, and 200-250% in hip surgery patients.

Overall Design and Plan of Study: 30 Surgical patients (type of elective surgery: total hip and total knee replacements) will be randomized into two arms of the study attempting to get a similar mean age for each group: Group 1: 15 patients receive placebo Day --8,--7,--6,--5,--4,--3,--2,--1,Day 0 (surgery), Post-op day 1,2,3, and 4. Group 2: 15 patients receive (10 mg) of Namenda (memantine) Day --8,--7,--6,--5,--4,--3,--2, then 20 mg per day on Day --1, day 0 (surgery), Post-op day 1,2,3 then 10 mg per day Post-op day 4, then stop Namenda.

Both groups will receive a MMSE, CLOX, Confusion Assessment Method (CAM) and the Delirium Rating Scale-Revised-98 Scale on day --8 (or before drug/placebo), day --1, then post-op day 1-6. Actigraphy will be performed day --8 through post-op day 6, and sleep diaries will be collected (subjected diaries pre-hospital day --8 through day --1, then objective diaries, day --1 through post-op day 6 in hospital).

Baseline screening blood tests will be drawn on all patients and include SMA-8 including BUN and creatinine, serum albumin, TSH, NH3 and baseline BP, Pulse and Temperature. Pre-op hematocrit has been shown to be a predictor as well, and may be worthwhile to follow up in these patients.

If delirium should develop in any patients, treatment will be as per usual standard of care, with likely psychiatric consultation and medications used will be tracked.

Pharmaco-economic arm (PEA) of syudy: We are working with hospital administration and will be able to obtain costs of care such as the following: room charges, locations (whether ICU, step-down unit or regular floor etc), pharmacy costs, cost of consultations needed, number of days in the hospital needed for each group. Discharge outcome (disposition, need for SNF vs. home, visiting nurse service needs) will be compared at discharge, and fo;;ow-up 30 days later.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable
* 50 years of age or older
* having elective joint replacement surgery or other orthopedic procedures that are major surgery and require general anesthesia.

Exclusion Criteria:

* Alcohol or sedative hypnotic abuse or dependence
* Pregnancy
* Dementia or MR/DD patients if they do not have sufficient capacity to understand the consent
* renal impairment or a creatinine of 1.4 or higher
* currently taking cholinesterase inhibitors.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-03; Study Completion 2006-09

PRIMARY OUTCOMES:
Incidence and severity of delirium measured by Delirium Rating Scale-Revised-98, MMSE. Confusion Assessment Method, Clock Drawing Tests (CLOX), DSM-IV-TR criteria for Delirium.

SECONDARY OUTCOMES:
Length and cost of stay, disposition, level of care required post hosptialization, hospitalization satisfaction, number of consultants involved, total costs of care.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Privitera, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Background] Schwartz TL, Masand PS. The role of atypical antipsychotics in the treatment of delirium. Psychosomatics. 2002 May-Jun;43(3):171-4. doi: 10.1176/appi.psy.43.3.171. PMID 12075031
- [Background] Breitbart W, Rosenfeld B, Roth A, Smith MJ, Cohen K, Passik S. The Memorial Delirium Assessment Scale. J Pain Symptom Manage. 1997 Mar;13(3):128-37. doi: 10.1016/s0885-3924(96)00316-8. PMID 9114631
- [Background] Bekker AY, Weeks EJ. Cognitive function after anaesthesia in the elderly. Best Pract Res Clin Anaesthesiol. 2003 Jun;17(2):259-72. doi: 10.1016/s1521-6896(03)00005-3. PMID 12817919
- [Background] Nishikawa K, Nakayama M, Omote K, Namiki A. Recovery characteristics and post-operative delirium after long-duration laparoscope-assisted surgery in elderly patients: propofol-based vs. sevoflurane-based anesthesia. Acta Anaesthesiol Scand. 2004 Feb;48(2):162-8. doi: 10.1111/j.0001-5172.2004.00264.x. PMID 14995937
- [Background] Inouye SK. Delirium in hospitalized elderly patients: recognition, evaluation, and management. Conn Med. 1993 May;57(5):309-15. No abstract available. PMID 8319447
- [Background] Inouye SK, Rushing JT, Foreman MD, Palmer RM, Pompei P. Does delirium contribute to poor hospital outcomes? A three-site epidemiologic study. J Gen Intern Med. 1998 Apr;13(4):234-42. doi: 10.1046/j.1525-1497.1998.00073.x. PMID 9565386
- [Background] McCusker J, Cole M, Abrahamowicz M, Primeau F, Belzile E. Delirium predicts 12-month mortality. Arch Intern Med. 2002 Feb 25;162(4):457-63. doi: 10.1001/archinte.162.4.457. PMID 11863480
- [Background] Inouye SK. Delirium in hospitalized older patients: recognition and risk factors. J Geriatr Psychiatry Neurol. 1998 Fall;11(3):118-25; discussion 157-8. doi: 10.1177/089198879801100302. PMID 9894730
- [Background] Breitbart W, Gibson C, Tremblay A. The delirium experience: delirium recall and delirium-related distress in hospitalized patients with cancer, their spouses/caregivers, and their nurses. Psychosomatics. 2002 May-Jun;43(3):183-94. doi: 10.1176/appi.psy.43.3.183. PMID 12075033
- [Background] Gustafson Y, Berggren D, Brannstrom B, Bucht G, Norberg A, Hansson LI, Winblad B. Acute confusional states in elderly patients treated for femoral neck fracture. J Am Geriatr Soc. 1988 Jun;36(6):525-30. doi: 10.1111/j.1532-5415.1988.tb04023.x. PMID 2897391
- [Background] Saravay SM, Strain JJ. APM Task Force on Funding Implications of Consultation-Liaison Outcome Studies. Special series introduction: a review of outcome studies. Psychosomatics. 1994 May-Jun;35(3):227-32. doi: 10.1016/S0033-3182(94)71771-0. No abstract available. PMID 8036252
- [Background] Thomas RI, Cameron DJ, Fahs MC. A prospective study of delirium and prolonged hospital stay. Exploratory study. Arch Gen Psychiatry. 1988 Oct;45(10):937-40. doi: 10.1001/archpsyc.1988.01800340065009. PMID 3138960
- [Background] Schor JD, Levkoff SE, Lipsitz LA, Reilly CH, Cleary PD, Rowe JW, Evans DA. Risk factors for delirium in hospitalized elderly. JAMA. 1992 Feb 12;267(6):827-31. PMID 1732655
- [Background] Cushman LA. Secondary neuropsychiatric complications in stroke: implications for acute care. Arch Phys Med Rehabil. 1988 Oct;69(10):877-9. PMID 3178456
- [Background] Kishi Y, Iwasaki Y, Takezawa K, Kurosawa H, Endo S. Delirium in critical care unit patients admitted through an emergency room. Gen Hosp Psychiatry. 1995 Sep;17(5):371-9. doi: 10.1016/0163-8343(95)00056-w. PMID 8522152
- [Background] Berggren D, Gustafson Y, Eriksson B, Bucht G, Hansson LI, Reiz S, Winblad B. Postoperative confusion after anesthesia in elderly patients with femoral neck fractures. Anesth Analg. 1987 Jun;66(6):497-504. PMID 3578861
- [Background] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384
- [Background] Foreman MD. Prevention and Treatment Strategies for Delirium. Primary Psychiatry 11(11): 52-58, 2004.
- [Background] Inouye SK, Bogardus ST Jr, Charpentier PA, Leo-Summers L, Acampora D, Holford TR, Cooney LM Jr. A multicomponent intervention to prevent delirium in hospitalized older patients. N Engl J Med. 1999 Mar 4;340(9):669-76. doi: 10.1056/NEJM199903043400901. PMID 10053175
- [Background] Bogardus ST Jr, Desai MM, Williams CS, Leo-Summers L, Acampora D, Inouye SK. The effects of a targeted multicomponent delirium intervention on postdischarge outcomes for hospitalized older adults. Am J Med. 2003 Apr 1;114(5):383-90. doi: 10.1016/s0002-9343(02)01569-3. PMID 12714128
- [Background] Rizzo JA, Bogardus ST Jr, Leo-Summers L, Williams CS, Acampora D, Inouye SK. Multicomponent targeted intervention to prevent delirium in hospitalized older patients: what is the economic value? Med Care. 2001 Jul;39(7):740-52. doi: 10.1097/00005650-200107000-00010. PMID 11458138
- [Background] Trzepacz PT. Delirium. Advances in diagnosis, pathophysiology, and treatment. Psychiatr Clin North Am. 1996 Sep;19(3):429-48. doi: 10.1016/s0193-953x(05)70299-9. PMID 8856810
- [Background] Kawashima T, Yamada S. Delirium caused by donepezil: a case study. J Clin Psychiatry. 2002 Mar;63(3):250-1. doi: 10.4088/jcp.v63n0312f. No abstract available. PMID 11926729
- [Background] Trzepacz PT. The neuropathogenesis of delirium. A need to focus our research. Psychosomatics. 1994 Jul-Aug;35(4):374-91. doi: 10.1016/S0033-3182(94)71759-X. PMID 7916159
- [Background] Rogawski MA. What is the rationale for new treatment strategies in Alzheimer's disease? CNS Spectr. 2004 Jul;9(7 Suppl 5):6-12. doi: 10.1017/s1092852900024743. PMID 15241294
- [Background] Nelson JK, Schilke DA. The evolution of psychiatric liaison nursing. Perspect Psychiatr Care. 1976 Apr-Jun;14(2):60-5. doi: 10.1111/j.1744-6163.1976.tb01536.x. No abstract available. PMID 1046580
- [Background] Chase TN. Levodopa therapy: consequences of the nonphysiologic replacement of dopamine. Neurology. 1998 May;50(5 Suppl 5):S17-25. doi: 10.1212/wnl.50.5_suppl_5.s17. PMID 9591518
- [Background] Harrell RG, Othmer E. Postcardiotomy confusion and sleep loss. J Clin Psychiatry. 1987 Nov;48(11):445-6. PMID 3680186
- [Background] Matsushima E, Nakajima K, Moriya H, Matsuura M, Motomiya T, Kojima T. A psychophysiological study of the development of delirium in coronary care units. Biol Psychiatry. 1997 Jun 15;41(12):1211-7. doi: 10.1016/s0006-3223(96)00219-3. PMID 9171911
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Trzepacz PT, Mittal D, Torres R, Kanary K, Norton J, Jimerson N. Validation of the Delirium Rating Scale-revised-98: comparison with the delirium rating scale and the cognitive test for delirium. J Neuropsychiatry Clin Neurosci. 2001 Spring;13(2):229-42. doi: 10.1176/jnp.13.2.229. PMID 11449030
- [Background] Gleason OC. Donepezil for postoperative delirium. Psychosomatics. 2003 Sep-Oct;44(5):437-8. doi: 10.1176/appi.psy.44.5.437. No abstract available. PMID 12954923
- [Background] Scarpini E, Scheltens P, Feldman H. Treatment of Alzheimer's disease: current status and new perspectives. Lancet Neurol. 2003 Sep;2(9):539-47. doi: 10.1016/s1474-4422(03)00502-7. PMID 12941576
- [Background] Wengel SP, Burke WJ, Roccaforte WH. Donepezil for postoperative delirium associated with Alzheimer's disease. J Am Geriatr Soc. 1999 Mar;47(3):379-80. doi: 10.1111/j.1532-5415.1999.tb03015.x. No abstract available. PMID 10078910
- [Background] Moster ML, Balcer LJ. The 56th annual meeting of the American Academy of Neurology, San Francisco, California, April 24-30, 2004. J Neuroophthalmol. 2004 Dec;24(4):327-36. doi: 10.1097/00041327-200412000-00012. No abstract available. PMID 15662251
- [Background] Rogawski MA, Wenk GL. The neuropharmacological basis for the use of memantine in the treatment of Alzheimer's disease. CNS Drug Rev. 2003 Fall;9(3):275-308. doi: 10.1111/j.1527-3458.2003.tb00254.x. PMID 14530799
- [Background] Cepeda C, Levine MS. Dopamine and N-methyl-D-aspartate receptor interactions in the neostriatum. Dev Neurosci. 1998;20(1):1-18. doi: 10.1159/000017294. PMID 9600386
- [Background] Cepeda C, Colwell CS, Itri JN, Gruen E, Levine MS. Dopaminergic modulation of early signs of excitotoxicity in visualized rat neostriatal neurons. Eur J Neurosci. 1998 Nov;10(11):3491-7. doi: 10.1046/j.1460-9568.1998.00357.x. PMID 9824462
- [Background] Huang KX, Bergstrom DA, Ruskin DN, Walters JR. N-methyl-D-aspartate receptor blockade attenuates D1 dopamine receptor modulation of neuronal activity in rat substantia nigra. Synapse. 1998 Sep;30(1):18-29. doi: 10.1002/(SICI)1098-2396(199809)30:13.0.CO;2-N. PMID 9704877
- [Background] Royall DR, Cordes JA, Polk M. CLOX: an executive clock drawing task. J Neurol Neurosurg Psychiatry. 1998 May;64(5):588-94. doi: 10.1136/jnnp.64.5.588. PMID 9598672
- [Background] Diagnostic and Statistical Manual of Mental Disorders, Forth Edition, Text Revision. Washington D.C., American Psychiatric Association, 2000.
- [Background] Cohen J. Statistical Power Analysis for the Behavioral Sciences, 2nd ed. Lawrence Erlbaum Associates, New Jersey.